CLINICAL TRIAL: NCT01775137
Title: A 48 Week Extension to CTBM100C2401, a Single Arm, Open-label, Multicenter, Phase IV Extension Trial to Assess Long Term Safety of Tobramycin Inhalation Powder (TIP) in Patients With Cystic Fibrosis Who Completed Participation in CTBM100C2401.
Brief Title: Ext. Long-term Safety Study in CF Patients: Single Arm TIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CTBM100C2401E1
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Long-term Safety of TIP
Keywords: CF, Open-label, TIP, phase IV, extension study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TBM100 (Experimental): TIP 112 mg/b.i.d
  Interventions: Drug: TBM100

INTERVENTIONS:
Drug: TBM100 — Tobramycin inhalation powder (TIP) 112mg/b.i.d

SUMMARY:
The purpose of this extension study is to collect additional 48 weeks of safety data from patients taking TIP who have completed the core study CTBM100C2401. The purpose of collecting second year safety data through this study is to obtain long-term (2 years) safety data of TIP.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the core study CTBM100C2401 and able to comply with all protocol requirements of the extension study

Exclusion Criteria:

* Serum creatinine 2mg/dl, BUN 40mg/dl or proteinuria 2+ or more at the time of entry into the extension
* Use of loop diuretics within 7 days prior to entry into the extension study
* Pregnant or nursing women
* Women of child bearing potential unless using highly effective method of contraception as indicated in the protoco

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (4):
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
- Argentina (3):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
- Australia (2):
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Budapest, Hungary
- Italy (5):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Palermo, Italy
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Roma
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 22 centers in 9 countries.
Pre-assignment Details: Of 96 participants who completed the core study (CTBM100C2401), NCT01519661; 45 participants were enrolled in the extension study.
Groups:
- Tobramycin Inhalation Powder: Participants inhaled four capsules of tobramycin inhalation powder (28 mg) twice daily (bid) via the T326 inhaler device, for 28 days (treatment phase in each cycle). Each treatment phase therefore consisted of 112 mg tobramycin (4 capsules of 28 mg each) with the total daily dose of 224 mg tobramycin (112 mg bid).The treatment phase was followed by 28 days of no study treatment (off treatment in each cycle). These 56 days represented 1 cycle of therapy.
Period: Overall Study
Arm/Group | Tobramycin Inhalation Powder
Started | 45
Completed | 34
Not Completed | 11
Not completed — Death | 1
Not completed — Protocol deviation | 2
Not completed — Unsatisfactory therapeutic effect | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by participants | 5

BASELINE CHARACTERISTICS:
Groups:
- Tobramycin Inhalation Powder: Participants inhaled four capsules of tobramycin inhalation powder (28 mg) bid via the T326 inhaler device, for 28 days (treatment phase in each cycle). Each treatment phase therefore consisted of 112 mg tobramycin (4 capsules of 28 mg each) with the total daily dose of 224 mg tobramycin (112 mg bid).The treatment phase was followed by 28 days of no study treatment (off treatment in each cycle). These 56 days represented 1 cycle of therapy.
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 33
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 25
Region of Enrollment [Number; unit: participants]
  Canada | 1
  Argentina | 9
  Hungary | 1
  United States | 6
  Italy | 7
  Mexico | 5
  Australia | 5
  Germany | 5
  Spain | 6
Pseudomonas aeruginosa tobramycin minimal inhibitory concentration (MIC) [Number; unit: Participants]
  > 8 microgram/milliliter(ug/mL) | 12
  <= 8 ug/mL | 33
Forced expiratory volume in one second (FEV1) percent (%) predicted [Mean (Standard Deviation); unit: Percent predicted] | 52.2 (15.01)
Forced vital capacity (FVC) % predicted [Mean (Standard Deviation); unit: Percent predicted] | 73.2 (17.49)
Forced expiratory flow from 25 to 75 % (FEF2575%) % predicted [Mean (Standard Deviation); unit: Percent predicted] | 24.7 (14.86)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), AEs/SAEs Leading to Discontinuation of Study Drug and Deaths Over 12 Treatment Cycles
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or encompassed any other clinically significant event that could jeopardize the participant or require medical or surgical intervention to prevent one of the aforementioned outcomes. Based on the severity, AEs were categorised into 3 types as mild, moderate and severe. Death was a fatal event leading to permanent cessations of all vital functions of the body.
Time Frame: Baseline (start of study treatment in core study) to Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population, defined as all the participants who entered the extension study and received at least one dose of study drug within the extension.
Measure: Number; unit: Participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Participants
  AEs | 39
  Mild AEs | 10
  Moderate AEs | 18
  Severe AEs | 11
  SAEs | 19
  Discontinued study drug due to AEs | 2
  Discontinued study drug due to SAEs | 1
  Deaths | 1

2. Secondary Outcome: Relative Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Percent Predicted Over 12 Treatment Cycles
Description: FEV1 was defined as the volume of air expired in 1 second. FEV1 was assessed as a pulmonary function by using spirometry tests in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) criteria. FEV1% predicted is a normalized value of FEV1 calculated using the Knudsen equation, based upon participant's age, gender and height. Relative change in FEV1 % predicted from baseline to pre-dose day X = ((pre-dose day*FEV1% predicted - baseline FEV1% predicted) / baseline FEV1 % predicted) x 100.
Time Frame: Baseline (start of study treatment in core study), Day 29, Day 85, Day 141, Day 197, Day 253, Day 309, Day 337, Day 365, Day 421, Day 477, Day 533, Day 589, Day 645, 673 (end of the extension study)
Population: Extension safety population, defined as all the participants who entered the extension study and received at least one dose of study drug within the extension and had FEV1% values at both baseline and the post baseline time points. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Percent change in FEV1 % predicted
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Percent change in FEV1 % predicted
  Core cycle 1, Day 29 (n=44) | 5.0 (20.36)
  Core cycle 2, day 85 (n=45) | 0.8 (19.51)
  Core cycle 3, day 141 (n=45) | 1.3 (15.32)
  Core cycle 4, day 197 (n=44) | 0.0 (17.34)
  Core cycle 5, day 253 (n=43) | -0.5 (17.91)
  Core cycle 6, day 309 (n=45) | -1.6 (14.19)
  Core study completion, (n=43) | -3.1 (19.72)
  Extension Cycle 7, day 337(n=44) | -5.2 (14.29)
  Extension Cycle 7, day 365(n=44) | -3.7 (14.84)
  Extension Cycle 8, day 421(n=41) | -6.1 (14.55)
  Extension Cycle 9, day 477(n=42) | -4.8 (14.03)
  Extension Cycle 10, day 533(n=39) | -7.5 (13.97)
  Extension Cycle 11, day 589(n=38) | -5.4 (19.49)
  Extension Cycle 12, day 645(n=35) | -7.5 (14.15)
  Extension completion, (n=33) | -9.3 (12.76)

3. Secondary Outcome: Absolute Change From Baseline in Pseudomonas Aeruginosa Sputum Density Over 12 Treatment Cycles
Description: Microbiological data was collected to understand the direct impact of the drug on the pathogens. Sputum samples were cultured for the presence of three Pseudomonas aeruginosa (P. aeruginosa) biotypes measured were mucoid, dry and small colony variant. Absolute change was determined using the formula = (Post-baseline value- baseline value). If no P. aeruginosa was isolated for a visit, log10 colony forming units (CFU) was imputed with log10 (19) for all biotypes.
Time Frame: Baseline (start of study treatment in core study), Day 29, Day 85, Day 141, Day 197, Day 253, Day 309, Day 337, Day
Measure: Mean (Standard Deviation); unit: log 10 CFU/g
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
log 10 CFU/g
  Core cycle 1, day 29 (n=42) | -1.9 (2.83)
  Core cycle 2, day 85 (n=43) | -1.5 (1.60)
  Core cycle 3, day 141 (n=44) | -1.4 (2.00)
  Core cycle 4, day 197 (n=41) | -1.2 (1.80)
  Core cycle 5, day 253 (n=40) | -2.2 (2.26)
  Core cycle 6, day 309 (n=39) | -1.4 (2.02)
  Core study completion, day 337 (n=42) | -0.7 (2.38)
  Extension cycle 7, day 337 (n=40) | -0.7 (2.46)
  Extension cycle 7, day 365 (n=41) | -1.4 (2.18)
  Extension cycle 8, day 421 (n=41) | -1.1 (2.20)
  Extension cycle 9, day 477 (n=39) | -1.1 (2.33)
  Extension cycle 10, day 533 (n=35) | -0.8 (1.97)
  Extension cycle 11, day 589 (n=36) | -1.0 (2.38)
  Extension cycle 12, day 645 (n=31) | -0.6 (1.96)
  Extension completion, day 673 (n=29) | -1.0 (2.70)

4. Secondary Outcome: Tobramycin Minimum Inhibitory Concentration (MIC) 50 and MIC 90 Values for Pseudomonas Aeruginosa Over 12 Treatment Cycles
Description: MIC was defined as the lowest concentration of an antimicrobial agent required to inhibit the visible growth of a microorganism after overnight incubation. Tobramycin MIC 50 and MIC 90 values were defined as the lowest concentration of tobramycin required to inhibit 50% and 90%, respectively, of the P. aeruginosa strains tested (mucoid,dry and small colony variant biotypes).
Time Frame: as for outcome 2
Population: The analysis was performed in extension safety population, who had microbiological data at specified time points. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Number; unit: micrograms/milliliters
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
micrograms/milliliters
  Core cycle, Baseline- MIC 50 (n=45) | 2
  Core cycle 1, day 29- MIC 50 (n=41) | 2
  Core cycle 2, day 85- MIC 50 (n=40) | 2
  Core cycle 3, day 141- MIC 50 (n=43) | 2
  Core cycle 4, day 197- MIC 50 (n=40) | 2
  Core cycle 5, day 253- MIC 50 (n=36) | 2
  Core cycle 6, day 309- MIC 50 (n=37) | 4
  Core study completion, Day 337- MIC 50 (n=40) | 2
  Extension cycle 7, day 337- MIC 50 (n=38) | 2
  Extension cycle 7, day 365- MIC 50 (n=38) | 2
  Extension cycle 8, day 421- MIC 50 (n=39) | 2
  Extension cycle 9, day 477- MIC 50 (n=39) | 4
  Extension cycle 10, day 533- MIC 50 (n=35) | 2
  Extension cycle 11, day 589- MIC 50 (n=36) | 2
  Extension cycle 12, day 645- MIC 50 (n=32) | 2
  Extension completion, Day 673 - MIC 50 (n=29) | 2
  Core cycle, Baseline- MIC 90 (n=45) | 32
  Core cycle 1, day 29- MIC 90 (n=41) | 256
  Core cycle 2, day 85- MIC 90 (n=40) | 256
  Core cycle 3, day 141- MIC 90 (n=43) | 512
  Core cycle 4, day 197- MIC 90 (n=40) | 128
  Core cycle 5, day 253- MIC 90 (n=36) | 256
  Core cycle 6, day 309- MIC 90 (n=37) | 512
  Core study completion, Day 337- MIC 90 (n=40) | 512
  Extension cycle 7, day 337- MIC 90 (n=38) | 512
  Extension cycle 7, day 365- MIC 90 (n=38) | 128
  Extension cycle 8, day 421- MIC 90 (n=39) | 128
  Extension cycle 9, day 477- MIC 90 (n=39) | 512
  Extension cycle 10, day 533- MIC 90 (n=35) | 256
  Extension cycle 11, day 589- MIC 90 (n=36) | 512
  Extension cycle 12, day 645- MIC 90 (n=32) | 512
  Extension completion, Day 673 - MIC 90 (n=29) | 512

5. Secondary Outcome: Percentage of Participants Who Used New Anti-pseudomonal Antibiotics Over 12 Treatment Cycles
Description: The rate of anti-pseudomonal antibiotics use were determined from the collection of concomitant medication during the study.
Time Frame: Baseline of core study, Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Percentage of participants | 77.8

6. Secondary Outcome: Total Number of Days of New Anti-pseudomonal Antibiotics Use Over 12 Treatment Cycles
Description: The total number of days with usage of new anti-pseudomonal antibiotic were determined.
Time Frame: Baseline of core study, Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Median (Full Range); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days
  Overall route (n=35) | 59.0 [15 to 252]
  Oral use (n=31) | 42.0 [11 to 175]
  i.v use (n=25) | 32.0 [7 to 252]
  Inhaled use (n=1) | 9.0 [9.0 to 9.0]

7. Secondary Outcome: Time to Use of New Anti-pseudomonal Antibiotics Over 12 Treatment Cycles
Description: Time to first usage of anti-pseudomonal antibiotic was determined using Kaplan Meier estimate. Participants without an event were censored at the date of the last available post-baseline measurement.
Time Frame: Baseline of core study, Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days | 202.0 [89.0 to 336.0]

8. Secondary Outcome: The Percentage of the Participants Hospitalized Due to Serious Respiratory-related AEs Were Determined During the Study.
Description: The percentage of the participants hospitalized due to serious respiratory-related AEs were determined during the study.
Time Frame: Baseline of core study, Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Percentage of participants | 40.0

9. Secondary Outcome: Number of Hospitalization Days Due to Respiratory Related Serious Adverse Events (SAEs) Over 12 Treatment Cycles
Description: The total number of hospitalization days due to serious respiratory-related adverse events was analyzed using Kaplan-Meier estimate.
Time Frame: Baseline of core study, Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population.
Measure: Median (Full Range); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days | 17.0 [4 to 129]

10. Secondary Outcome: Time to First Hospitalization Due to Respiratory Related Serious Adverse Events (SAEs) Over 12 Treatment Cycles
Description: The day of first hospitalization due to serious respiratory-related adverse events was analysed using Kaplan Meier estimate.
Time Frame: Baseline of core study, Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days | NA [NA to NA] — Here, value is not applicable due to insufficient number of events.

11. Secondary Outcome: Acute Relative Change From Pre-dose to 30-minute Post-dose in Forced Expiratory Volume in One Second (FEV1) Percent Predicted Over 12 Treatment Cycles
Description: FEV1 was defined as the volume of air expired in 1 second. FEV1 was assessed as a pulmonary function by using spirometry tests in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) criteria. Relative change in FEV1 % predicted was calculated by using the formula = 100 *(30-min post-dose value - pre-dose value) / pre-dose value.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent change in FEV1 % predicted
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Percent change in FEV1 % predicted
  Core cycle 1, day 1 (n=44) | -4.9 (6.72)
  Core cycle 1, day 29 (n=41) | -3.5 (4.25)
  Core cycle 2, day 85 (n=39) | -3.5 (6.19)
  Core cycle 3, day 141 (n=42) | -2.6 (6.06)
  Core cycle 4, day 197 (n=40) | -3.2 (5.41)
  Core cycle 5, day 253 (n=41) | -3.8 (5.47)
  Core cycle 6, day 309 (n=39) | -2.5 (5.94)
  Extension cycle 7, day 365(n=37) | -0.1 (7.79)
  Extension cycle 8, day 421(n=36) | -3.7 (5.10)
  Extension cycle 9, day 477(n=37) | -3.5 (4.78)
  Extension cycle 10, day 533(n=36) | -1.0 (12.54)
  Extension cycle 11, day 589(n=35) | -3.3 (6.73)
  Extension cycle 12, day 645(n=30) | -3.1 (4.01)

12. Secondary Outcome: Relative Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Percent Predicted Over 6 Treatment Cycles in Extension Study
Description: as for outcome 2
Time Frame: Baseline (start of study treatment in extension study), Day 365, Day 421, Day 477, Day 533, Day 589, Day 645, 673 (end of the extension study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change in FEV1 % predicted
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Percent change in FEV1 % predicted
  Extension Cycle 7, day 365(n=44) | 4.0 (16.93)
  Extension Cycle 8, day 421(n=41) | 2.4 (13.71)
  Extension Cycle 9, day 477(n=42) | 2.4 (16.18)
  Extension Cycle 10, day 533(n=39) | -1.4 (13.75)
  Extension Cycle 11, day 589(n=38) | 0.3 (14.76)
  Extension Cycle 12, day 645(n=35) | -0.6 (13.95)
  Extension completion, (n=33) | -3.5 (10.74)

13. Secondary Outcome: Absolute Change From Baseline in Pseudomonas Aeruginosa Density Over 6 Treatment Cycles in Extension Study
Description: Microbiological data was collected to understand the direct impact of the drug on the pathogens. Sputum samples were cultured for the presence of three Pseudomonas aeruginosa (P. aeruginosa) biotypes measured were mucoid, dry and small colony variant. If no P. aeruginosa was isolated for a visit, log10 colony forming units (CFU) was imputed with log10 (19) for all biotypes. Absolute change was calculated by using the formula = (Value at actual time point - start of extension value).
Time Frame: as for outcome 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 CFU
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
log10 CFU
  Extension Cycle 7, day 365(n=38) | -0.7 (2.77)
  Extension Cycle 8, day 421(n=39) | -0.2 (2.60)
  Extension Cycle 9, day 477(n=39) | -0.2 (2.51)
  Extension Cycle 10, day 533(n=35) | 0.2 (2.89)
  Extension Cycle 11, day 589(n=36) | 0.0 (2.49)
  Extension Cycle 12, day 645(n=32) | 0.4 (2.75)
  Extension completion, (n=29) | 0.3 (2.48)

14. Secondary Outcome: Percentage of Participants Who Used New Anti-pseudomonal Antibiotics in Extension Study
Description: as for outcome 5
Time Frame: Baseline of extension study, Day 673 (end of extension study)
Population: The analysis was performed in extension safety population.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Percentage of participants | 68.9

15. Secondary Outcome: Total Number of Days of New Anti-pseudomonal Antibiotics Use in Extension Study
Description: The total number of days with usage of new anti-pseudomonal antibiotic were determined.
Time Frame: Baseline of extension study, Day 673 (end of extension study)
Population: The analysis was performed in extension safety population.The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively
Measure: Median (Full Range); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days
  Overall route (n=31) | 33.0 [1 to 252]
  Oral use (n=23) | 28.0 [1 to 44]
  i.v use (n=20) | 16.0 [7 to 252]
  Inhaled use (n=1) | 9.0 [9 to 9]

16. Secondary Outcome: Time to Use of New Anti-pseudomonal Antibiotics in Extension Study
Description: as for outcome 7
Time Frame: Baseline of extension study, Day 673 (end of extension study)
Population: The analysis was performed in extension safety population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days | 139 [86 to 271]

17. Secondary Outcome: Percentage of Participants Hospitalized Due to Respiratory Related Serious Adverse Events (SAEs) in Extension Study
Description: The percentage of the participants hospitalized due to serious respiratory-related AEs were determined during the extension study.
Time Frame: Baseline of extension study, Day 673 (end of the extension study)
Population: The analysis was performed in extension safety population.
Measure: Number; unit: Percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Percentage of participants | 35.6

18. Secondary Outcome: Number of Hospitalization Days Due to Respiratory Related Serious Adverse Events (SAEs) in Extension Study
Description: The total number of hospitalisation days due to serious respiratory-related adverse events was analysed using Kaplan-Meier estimate.
Time Frame: Baseline of extension study, Day 673 (end of extension study)
Population: The analysis was performed in extension safety population.
Measure: Median (Full Range); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days | 16.0 [5 to 64]

19. Secondary Outcome: Time to First Hospitalization Due to Respiratory Related Serious Adverse Events (SAEs) in Extension Study
Description: The day of first hospitalization due to serious respiratory related adverse events was analysed using Kaplan Meier estimate.
Time Frame: Baseline of extension study, Day 673 (end of extension study)
Population: The analysis was performed in extension safety population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Days | NA [NA to NA] — Here, value is not applicable due to insufficient number of events.

20. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), AEs/SAEs Leading to Discontinuation of Study Drug and Deaths Over 6 Treatment Cycles in Extension Study
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalisation, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or encompassed any other clinically significant event that could jeopardize the participant or require medical or surgical intervention to prevent one of the aforementioned outcomes. Death was a fatal event leading to permanent cessations of all vital functions of the body.
Time Frame: Baseline (start of study treatment in extension study) to Day 673 (end of the extension study)
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 45
Number of participants
  AEs | 36
  SAEs | 16
  Discontinued study drug due to AEs | 1
  Discontinued study drug due to SAEs | 0
  Deaths | 1

ADVERSE EVENTS:
Time Frame: Baseline (start of study treatment in extension study) to Day 673 (end of the extension study)
Groups:
- Core: Eligible participants were assigned to four capsules of TIP at 28 mg dosage strength, inhaled b.i.d. in the morning and in the evening via the T-326 inhaler, for 28 days (on treatment), followed by 28 days of no study treatment (off treatment). Each treatment therefore consisted of 112 mg tobramycin (4 capsules of 28 mg each) with the total daily dose = 224 mg tobramycin (112 mg b.i.d.). These 56 days represented 1 cycle of therapy during core study.
- Extension: Participants inhaled four capsules of tobramycin inhalation powder (28 mg) bid via the T-326 inhaler device, for 28 days (treatment phase in each cycle). Each treatment phase therefore consisted of 112 mg tobramycin (4 capsules of 28 mg each) with the total daily dose of 224 mg tobramycin (112 mg bid). The treatment phase was followed by 28 days of no study treatment (off treatment in each cycle). These 56 days represented 1 cycle of therapy.
- Overall: All participants who inhaled tobramycin inhalation powder during both core and extension study.
Arm/Group | Core | Extension | Overall
Serious Adverse Events (participants affected / at risk) | 12/45 | 16/45 | 19/45
Other Adverse Events (participants affected / at risk) | 33/45 | 32/45 | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core (N=45) | Extension (N=45) | Overall (N=45)
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 11 | 14 | 17
Influenza (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Forced expiratory volume decreased (Investigations) | 0 | 1 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Haemodynamic instability (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core (N=45) | Extension (N=45) | Overall (N=45)
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 7
Constipation (Gastrointestinal disorders) | 0 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Chest discomfort (General disorders) | 1 | 2 | 2
Fatigue (General disorders) | 2 | 3 | 4
Pyrexia (General disorders) | 3 | 2 | 4
Bacterial disease carrier (Infections and infestations) | 1 | 3 | 3
Ear infection (Infections and infestations) | 2 | 0 | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 18 | 16 | 25
Nasopharyngitis (Infections and infestations) | 9 | 9 | 13
Pharyngitis (Infections and infestations) | 2 | 0 | 2
Rhinitis (Infections and infestations) | 2 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Forced expiratory volume decreased (Investigations) | 4 | 5 | 8
Pulmonary function test decreased (Investigations) | 2 | 0 | 2
Staphylococcus test positive (Investigations) | 3 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 4 | 4 | 6
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hypertension (Vascular disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e, data from all sites) in the clinical trial.